CLINICAL TRIAL: NCT07257653
Title: The Safety and Efficacy of Cetuximab Beta Plus Fruquintinib With or Without Immune Checkpoint Inhibitorrs in First-line Treatment of RAS/BRAF Wild Type Unresectable Metastatic Colorectal Cancer
Acronym: concept
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Ding Ke-Feng, Professor, Second Affiliated Hospital, School of Medicine, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: concept
Record Dates: First submitted 2025-11-20; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Colorectal Neoplasms; RAS; BRAF; Cetuximabβ; Fruquintinib
Keywords: Colorectal cancer; Chemotherapy-free; KRAS/NRAS/BRAF wild-type; cetuximab combined with fruquintinib; with or without immune checkpoint inhibitors
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Arm A: Cetuximab β + Fruquintinib Arm B: Cetuximab β + Fruquintinib + anti-PD1 antibody Arm C: Cetuximab β + Fruquintinib + anti-PD1/CTLA4 antibody
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm A (Experimental): Cetuximab β + Fruquintinib
  Interventions: Drug: Cetuximab β；Fruquintinib；
- Arm B (Experimental): Cetuximab β + Fruquintinib + anti-PD1 antibody
  Interventions: Drug: Cetuximab β；Fruquintinib；anti-PD1 antibody；
- Arm C (Experimental): Cetuximab β + Fruquintinib + anti-PD1/CTLA4 antibody
  Interventions: Drug: Cetuximab β；Fruquintinib；anti-PD1/CTLA4 antibody

INTERVENTIONS:
Drug: Cetuximab β；Fruquintinib； — Arm A：Cetuximab β（500mg/m2,iv,d1,q2w）+Fruquintinib(5mg, po, qd, 2w/1w)；
  Arms: Arm A
Drug: Cetuximab β；Fruquintinib；anti-PD1 antibody； — Arm B：Cetuximab β (500mg/m2,iv,d1,q2w）+Fruquintinib（5mg, po, qd, 2w/1w）+Sintilimab（200mg, iv, d1, q3w）；
  Arms: Arm B
Drug: Cetuximab β；Fruquintinib；anti-PD1/CTLA4 antibody — Arm C：Cetuximab β(500mg/m2,iv,d1,q2w）+Fruquintinib（5mg, po, qd, 2w/1w）+anti-PD1/CTLA4 antibody(5mg/kg, d1, q3w)
  Arms: Arm C

SUMMARY:
Colorectal cancer is a malignant tumor ranking among the top four in incidence and the top three in causes of death globally . Chemotherapy combined with anti-EGFR or anti-VEGF monoclonal antibodies is currently the standard first-line treatment for advanced pMMR colorectal cancer. The inclusion of anti-EGFR or anti-VEGF targeted therapies has improved the overall survival of advanced colorectal cancer patients from 13 months in the era of fluorouracil monotherapy to the current 30 months.

However, many patients refuse chemotherapy or cannot tolerate cytotoxic chemotherapeutic drugs, which often leads to poor prognosis in advanced colorectal cancer. Thus, in the treatment of advanced colorectal cancer, is it possible to achieve antitumor activity through the combination of targeted drugs while avoiding chemotherapy?

Early clinical studies evaluated the possibility of combining anti-EGFR and anti-VEGF monoclonal antibodies. Subsequent large-scale Phase III clinical studies, such as PACCE , indicated that the combination of FOLFOX or FOLFIRI regimens with bevacizumab and panitumumab increased adverse reactions without providing survival benefits in the overall colorectal cancer population compared to the control group. Following this, the CAIRO2 clinical study added cetuximab to CapeOX combined with bevacizumab and still did not demonstrate survival benefits in the first-line treatment of advanced colorectal cancer, particularly in patients with RAS mutations. However, subgroup analyses suggested a certain survival advantage in patients with wild-type RAS who received combined targeted therapy. A recent clinical study (ECOG-ACRIN E7208) showed that in patients with KRAS wild-type advanced colorectal cancer, second-line use of irinotecan combined with cetuximab and ramucirumab significantly improved progression-free survival (PFS) and disease control rate (DCR) compared to cetuximab combined with irinotecan. These studies suggest that combining anti-EGFR and anti-VEGF monoclonal antibodies is a feasible approach for patients with wild-type RAS

Certainly, in terms of anti-VEGF options, besides macromolecular anti-VEGFR monoclonal antibodies, small-molecule tyrosine kinase inhibitors targeting VEGF have also demonstrated significant antitumor activity in colorectal cancer. Studies have shown that fruquintinib significantly prolongs the survival of patients with advanced colorectal cancer, leading to its approval as a third-line treatment for colorectal cancer.

On the other hand, immunotherapy targeting PD-1 and CTLA-4 has recently made significant progress in the treatment of colorectal cancer. For the pMMR type, which accounts for over 90% of advanced colorectal cancer cases, related clinical studies have confirmed that the combination of immunotherapy and targeted therapy has significant antitumor synergistic effects. These studies also indicate that immune checkpoint inhibitors can enhance the antitumor activity of anti-EGFR and anti-VEGF targeted therapies in pMMR advanced colorectal cancer.

This study aims to evaluate the efficacy and safety of cetuximab combined with fruquintinib, with or without immune checkpoint inhibitors, as a first-line treatment for pMMR, RAS/BRAF wild-type metastatic colorectal cancer.

DETAILED DESCRIPTION:
According to the study design, 90 patients aged 18 to 80 years, with an ECOG score of 0-1, histologically confirmed colorectal adenocarcinoma, pMMR, KRAS/NRAS/BRAF wild-type, and unresectable metastases, including at least one measurable lesion as per RECIST 1.1 criteria, will be randomly assigned to three groups. They will receive the following treatments:

Arm A: Cetuximab β + Fruquintinib Arm B: Cetuximab β + Fruquintinib + anti-PD1 antibody Arm C: Cetuximab β + Fruquintinib + anti-PD1/CTLA4 antibody The primary endpoint is progression-free survival (PFS), and secondary endpoints include safety, ORR, and DCR.

ELIGIBILITY:
Inclusion Criteria:

1）Subjects voluntarily join this study, sign the informed consent form, and demonstrate good compliance; 2) Age: 10-80 years old, ECOG PS score of 0-1. For patients aged 80-85, comprehensive functional assessments must be completed, and they may be enrolled if the investigator deems them tolerable, with an expected survival of over 3 months; 3) Histopathologically and/or cytologically confirmed, unresectable metastatic colorectal adenocarcinoma confirmed by MDT discussion (UICC/AJCC TNM staging system for colorectal cancer, 8th Edition, 2017); 4) At least one measurable lesion confirmed according to RECIST 1.1 criteria; 5) Adequate function of major organs, meeting the following criteria:

1. Hematological examination standards (no blood transfusion or use of hematopoietic growth factors for correction within 7 days prior to screening):

   1. Hemoglobin (HGB) ≥ 90 g/L;
   2. Absolute neutrophil count (NEUT) ≥ 1.5 × 10⁹/L;
   3. Platelet count (PLT) ≥ 75 × 10⁹/L;
2. Biochemical tests must meet the following criteria:

   1. Total bilirubin (TBIL) ≤ 1.5 × ULN (≤ 3 × ULN for subjects with Gilbert's syndrome);
   2. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN. If with liver metastases, ALT and AST ≤ 5 × ULN;
   3. Serum creatinine (CR) ≤ 1.5 × ULN or creatinine clearance rate (CCR) ≥ 50 ml/min.
3. Coagulation function or thyroid function tests must meet the following criteria:

   1. Prothrombin time (PT), activated partial thromboplastin time (APTT), international normalized ratio (INR) ≤ 1.5 × ULN (without anticoagulant therapy);
   2. Thyroid-stimulating hormone (TSH) ≤ ULN; if abnormal, T3 and T4 levels should be assessed (FT3 and FT4 may be substituted if T3/T4 are unavailable at the center). Subjects may be enrolled if T3 and T4 levels are normal.
4. Echocardiogram assessment: Left ventricular ejection fraction (LVEF) ≥ 50%.
5. Hepatitis B surface antigen (HBsAg) negative. If HBsAg positive, hepatitis B virus deoxyribonucleic acid (HBV-DNA) must be < 2500 copies/mL or 500 IU/mL for enrollment.
6. HCV antibody negative or HCV-RNA negative subjects may enroll; if HCV-RNA positive, subjects must have alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 × ULN to enroll. Subjects with co-infection of hepatitis B and hepatitis C are excluded (positive for HBsAg or HBcAb, and positive for HCV antibody).
7. Female patients must meet one of the following conditions:

   1. Postmenopausal (defined as no menses for at least 1 year, with no other confirmed causes besides menopause), or
   2. Surgically sterilized (removal of ovaries and/or uterus), or
   3. Of childbearing potential but must meet the following:

      * Serum/urine pregnancy test within 7 days prior to enrollment must be negative;
      * Agree to use contraception with a failure rate of < 1% per year or maintain abstinence (avoiding heterosexual intercourse) (from signing the ICF until at least 6 months after the last dose of the study drug) (contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, correct use of hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, copper intrauterine devices, or condoms);
      * Must not be breastfeeding.
8. Male patients must meet the following: Agree to abstinence (avoiding heterosexual intercourse) or use contraception, as specified: When the partner is a woman of childbearing potential or is pregnant, the male patient must remain abstinent or use a condom during the treatment period and for at least 6 months after the last dose to prevent fetal drug exposure. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or post-ovulation methods) and withdrawal are not acceptable methods of contraception.

Exclusion Criteria:

1. Presence of MSI-H/dMMR patients.
2. Concurrent diseases and medical history:

   1. Diagnosis of or concurrent other malignancies within the past 3 years. The following conditions are eligible for enrollment:

      Cured cervical carcinoma in situ, non-melanoma skin cancer, and superficial bladder tumors [Ta (non-invasive tumor), Tis (carcinoma in situ), and T1 (tumor invading the basement membrane)];
   2. Multiple factors affecting oral medication (e.g., inability to swallow, chronic diarrhea, intestinal obstruction, etc.);
   3. History or tendency of gastrointestinal bleeding or perforation within 4 weeks prior to enrollment;
   4. Patients with active inflammatory bowel disease within 4 weeks prior to enrollment;
   5. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage;
   6. Unresolved toxicities from any prior antitumor therapy exceeding CTCAE Grade 1 (excluding alopecia and oxaliplatin-induced neurotoxicity ≤ Grade 2);
   7. Major surgical treatment, incisional biopsy, or significant traumatic injury within 28 days prior to the start of study treatment (excluding gastrointestinal endoscopic biopsy);
   8. Symptoms of active bleeding within 1 week prior to screening, without significant improvement or control;
   9. Patients with any bleeding event ≥ CTCAE Grade 3 within 4 weeks prior to study initiation, or presence of unhealed wounds, ulcers, or fractures;
   10. Arterial/venous thrombotic events within 6 months, such as cerebrovascular accidents (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis, and pulmonary embolism;
   11. History of psychoactive drug abuse with inability to abstain;
   12. Patients with any severe and/or uncontrolled diseases, including:

       * Uncontrolled hypertension (systolic blood pressure ≥150 mmHg or diastolic blood pressure ≥100 mmHg after standard antihypertensive therapy);
       * Myocardial ischemia ≥ Grade 2, myocardial infarction, arrhythmias (including QTc ≥450 ms for males, QTc ≥470 ms for females), and congestive heart failure ≥ Grade 2 (New York Heart Association (NYHA) classification);
       * Active or uncontrolled severe infections (≥ CTCAE Grade 2 infection);
       * Liver cirrhosis, active hepatitis*; (*Active hepatitis [Hepatitis B reference: HBsAg positive and HBV DNA positive (>2500 copies/mL or >500 IU/mL); Hepatitis C reference: HCV antibody positive and HCV viral titer above the upper limit of normal]. Note: Eligible HBsAg-positive or HBcAb-positive subjects and hepatitis C patients require continuous antiviral therapy to prevent viral reactivation.)
       * Renal failure requiring hemodialysis or peritoneal dialysis;
       * History of immunodeficiency, including HIV positivity or other acquired or congenital immunodeficiency diseases, or history of organ transplantation;
       * Poorly controlled diabetes (fasting blood glucose >10 mmol/L);
       * Urinalysis showing urine protein ≥++ and confirmed 24-hour urine protein quantification >1.0 g;
       * History of clear neurological or psychiatric disorders, including epilepsy or dementia requiring treatment.
   13. Patients with known active or suspected autoimmune diseases. Patients with immune-related hypothyroidism requiring thyroid hormone replacement therapy and well-controlled type I diabetes are allowed. Patients with vitiligo requiring no intervention or resolved childhood asthma/allergies requiring no intervention in adulthood are allowed.

       * Receipt of live vaccines within 28 days prior to enrollment. However, inactivated viral vaccines for seasonal influenza are permitted, while live attenuated influenza vaccines administered intranasally are not allowed.
       * Patients requiring systemic glucocorticoids (>10 mg/day prednisone equivalent) or other immunosuppressive drugs within 14 days prior to enrollment or during the study. The following conditions are allowed for enrollment:
       * Use of topical or inhaled glucocorticoids in the absence of active autoimmune diseases;
       * Adrenal glucocorticoid replacement therapy at doses ≤10 mg/day prednisone equivalent.
   14. Participation in other clinical studies or initiation of study treatment within 14 days after the end of prior clinical study treatment. History of severe allergy to any monoclonal antibody.
3. Tumor-related symptoms and treatment:

   1. Surgery (excluding prior diagnostic biopsies), radiotherapy, chemotherapy, or other anticancer therapies within 4 weeks prior to the start of study treatment (calculated from the end date of the last treatment as the washout period);
   2. Prior postoperative adjuvant therapy containing anti-angiogenic targeted drugs (including bevacizumab, cetuximab, panitumumab, aflibercept, regorafenib, etc.);

   d) Patients with symptomatic brain metastases or those whose symptoms have been controlled for less than 2 months;
4. Patients deemed by the investigator to have concomitant diseases that seriously endanger subject safety or affect study completion, or who are otherwise considered unsuitable for enrollment.

Ages: 10 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-10-21 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
PFS | 1 year
  PFS refers to the time from randomization (or the start of treatment) until the first observation of disease progression or death from any cause. The analysis is based on the full analysis set and the per-protocol set. The median PFS and its 95% CI were estimated using the Kaplan-Meier method, and survival curves were plotted.

SECONDARY OUTCOMES:
OS | 2 years
  OS refers to the time from randomization until death from any cause. The analysis is based on the full analysis set and the per-protocol set. The median OS and its 95% CI were estimated using the Kaplan-Meier method, and survival curves were plotted.
ORR | 1 year
  ORR：The proportion of patients in a study who have achieved a predefined reduction in tumor burden for a minimum period of time. This includes patients with either a Complete Response (CR) or a Partial Response (PR)
DCR | 1 year
  DCR：The proportion of patients in a study who have achieved Objective Response (CR or PR) or Stable Disease (SD) for a minimum specified duration.
DOR | 1 year
  DOR：The time from when Objective Response (CR or PR) is first documented to the time of disease progression or death from any cause, whichever occurs first. This metric is calculated only for patients who have achieved an objective response.

CONTACTS AND LOCATIONS:
Overall Officials: Kefeng Ding, PhD, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- Second Affiliated Hospital Zhejiang University College of Medicine, Hangzhou, Zhejiang Province 310999, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No